CLINICAL TRIAL: NCT03002220
Title: A Phase II Clinical Trial of Radium-223 Activity in Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC) With Asymptomatic Progression While on Abiraterone Acetate or Enzalutamide Besides AR-V7 Mutational Status
Brief Title: Trial of Rad-223 Activity in Asymptomatic Patients With mCRPC While on Abiraterone or Enzalutamide Besides AR-V7 Status
Acronym: EXCAAPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP098; 2016-001888-36 (EudraCT Number)
Record Dates: First submitted 2016-10-20; First posted 2016-12-23 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open-label (Experimental): Patient will be treated with radium-223 at a dose of 55 kilobecquerel (kBq) (after 2015 National Institute of Standards and Technology's (NIST) implementation) per kilogram body weight, given at four-week intervals for six intravenous injections.
  Interventions: Drug: radium-223

INTERVENTIONS:
Drug: radium-223 — Radium-223 at a dose of 55 kBq
  Other Names: Xofigo

SUMMARY:
Radium-223 is indicated for the treatment of patients with mCRPC with symptomatic bone metastases and no known visceral metastatic disease. However, very few data have been reported in patients with mCRPC who are asymptomatic or mildly symptomatic. Recently, results from an International Expanded Access Program have also suggested a benefit of radium-223 in asymptomatic patients with mCRPC. In addition, the mechanism of action of radium-223 should not be correlated with the presence/absence of the AR-V7 mutation, although this issue has not yet been evaluated.

The aim of this study is to assess the efficacy of radium-223 in asymptomatic patients with mCRPC, and to establish the association between AR-V7 status and radium-223 activity.

DETAILED DESCRIPTION:
Primary objective:

To assess the efficacy of radium-223 in asymptomatic patients with mCRPC who have progressed while on abiraterone acetate or enzalutamide treatment.

Primary endpoint:

To determine the efficacy of radium-223 in terms of radiological rPFS.

Secondary objectives:

* Safety profile.
* To determine the association between AR-V7 status (positive vs. negative) and PFS.
* To establish the relationship between CTCs number with radium-223 efficacy.

Secondary endpoints:

Safety AEs will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) of the US National Cancer Institute (NCI) version 4.0 [20]. Grade 3 or 4 AEs and serious adverse events (SAEs) will be assessed to determine the safety and tolerability of the various combinations of drugs.

Efficacy

* Radiographic progression-free survival (rPFS) depending on AR-V7 status.
* Overall survival (OS).
* Time to first symptomatic skeletal event (SSE).
* Time to prostate specific antigen (PSA) progression according to the Alpharadin in Symptomatic Prostate Cancer (ALSYMPCA) study criteria.
* Determination percentage of PSA progression.
* Alkaline phosphatase level response (AF), normalization of alkaline phosphatase level, according to the ALSYMPCA study criteria.

Molecular aspects

* Assessment of AR-V7 mutation evolution during the study treatment.
* Determination changes in CTCs number during the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult ≥ 18 years at the time of informed consent and has signed informed consent before any trial related activities and according to local guidelines.
* Subject has histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.
* Subject has bone metastases due to the prostate cancer and absence of visceral metastases.
* Subject has a serum testosterone of ≤ 1.7 nmol/L (or ≤ 50 ng/dL) at screening.
* Subject must have received a minimum of 24 weeks of treatment with abiraterone acetate or enzalutamide within its approved label indication and has discontinued use at least four weeks prior to start of study drug at day 1.
* Prior use of docetaxel is allowed in castration-naïve patients (maximum of six cycles).
* Subject receives and will continue to receive ongoing androgen deprivation with luteinising hormone-releasing hormone (LHRH) analogue therapy throughout the course of the study or has had a bilateral orchiectomy.
* Subject is asymptomatic from prostate cancer, defined as patients with the score on brief pain inventory (short form) (BPI-SF) Question #3 must zero and no use of opiate analgesics for prostate cancer-related pain currently or anytime within two weeks prior to screening.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at screening.
* Subject receiving bisphosphonate or other approved bone-targeting therapy must have been on stable doses for at least four weeks prior to start of study drug at day 1.
* Subject has a life expectancy of more than or equal to 12 months.
* Subject agrees not to participate in another interventional study while on study drug.
* Subject and his female partner who is of childbearing potential must use two acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for six months after final study drug administration.

Exclusion Criteria:

* Subject has received any anti-neoplastic therapy (including ketoconazole and chemotherapy) following abiraterone acetate or enzalutamide discontinuation and prior to start of study drug at day 1.
* Subject has known or suspected brain metastases or active leptomeningeal disease.
* Subject has concurrent disease or any clinically significant abnormality following the investigator's review of the physical examination and safety laboratory tests at screening, which in the judgment of the investigator would interfere with the subject's participation in this study or evaluation of study results.
* Subject has a history of another invasive cancer within three years prior to screening, with the exceptions of non-melanoma skin cancers or a non-infiltrating muscle bladder cancer that have a remote probability of recurrence in the opinion of the investigator in consultation with the medical monitor.
* Subject had major surgery within one month prior to screening.
* Subject has received investigational therapy within 28 days or 5 half lives, whichever is longer, prior to start of study drug at day 1.
* Subject has absolute neutrophil count < 1,500/μL, platelet count < 100,000/μL, and hemoglobin < 6.25 mmol/L (or < 10 g/dL) at screening (Note: Subjects must not have received any growth factors or blood transfusions within seven days of the hematologic laboratory values obtained at screening).
* Subject has total bilirubin > 1.5 times the upper limit of normal (ULN) at screening, except for subjects with documented Gilbert's syndrome.
* Subject has creatinine > 2.5 mg/dL at screening.
* Subject has albumin ≤ 30 g/L (or ≤ 3.0 g/dL) at screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Carles Galcerán, Study Director — H. Vall Hebrón
Locations (6):
- Spain (6):
  - MedSIR Investigative site, Barcelona
  - MedSIR Investigative site, Cáceres
  - MedSIR Investigative site, Córdoba
  - MedSIR Investigative site, Lugo
  - MedSIR Investigative site, Madrid
  - MedSIR investigative site, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carles J, Alonso-Gordoa T, Mellado B, Mendez-Vidal MJ, Vazquez S, Gonzalez-Del-Alba A, Piulats JM, Borrega P, Gallardo E, Morales-Barrera R, Paredes P, Reig O, Garcias de Espana C, Collado R, Bonfill T, Suarez C, Sampayo-Cordero M, Malfettone A, Garde J. Radium-223 for patients with metastatic castration-resistant prostate cancer with asymptomatic bone metastases progressing on first-line abiraterone acetate or enzalutamide: A single-arm phase II trial. Eur J Cancer. 2022 Sep;173:317-326. doi: 10.1016/j.ejca.2022.06.057. Epub 2022 Aug 16. PMID 35981452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2016 (first patient in) and October 2018, 52 (82.5%) men from 63 patients with mCRPC with asymptomatic progression while on abiraterone acetate or enzalutamide were included in the study from 9 sites in Spain.
  In the protocol, the information stating that the trial would start in November was mostly an approximation. However, the trial ended up starting the following month.
Pre-assignment Details: Men ≥ 18 years. Signed ICF. mCRPC with bone metastases and asymptomatic progression. Serum testosterone levels ≤ 1.7 nmol/L at screening. Minimum of 24 weeks of treatment with abiraterone acetate or enzalutamide. Ongoing androgen deprivation with luteinizing releasing hormone (LHRH) analogue therapy or bilateral orchiectomy. ECOG score ≤ 1. Life expectancy ≥ 12w. Subject with female partner who is of childbearing potential must use two acceptable methods of birth control.
Groups:
- Open-label: Patient will be treated with radium-223 at a dose of 55 kBq (after 2015 NIST implementation) per kilogram body weight, given at four-week intervals for six intravenous injections.
  radium-223: Radium-223 at a dose of 55 kBq
Period: Overall Study
Arm/Group | Open-label
Started | 52
Completed | 31
Not Completed | 21
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Disease progression | 13
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 52
Age, Continuous [Median (Full Range); unit: years] | 76.1 [69.4 to 82.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 52
Region of Enrollment [Number; unit: participants]
  Spain | 52

OUTCOME MEASURES:

1. Primary Outcome: Assess the Efficacy of Radium-223 in Terms of Radiological rPFS
Description: The primary efficacy endpoint is the median PFS (evaluated using RECIST v1.1) achieved with radium-223 treatment
Time Frame: From date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-label
Number analyzed (Participants) | 52
months | 5.53 [5.3 to 5.6]

2. Secondary Outcome: AEs and Serious Adverse Events (SAEs)
Time Frame: Starting from the first procedure required by the study up to three months after study discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 52
Participants | 46

3. Secondary Outcome: Radiographic Progression-free Survival (rPFS) Depending on AR-V7 Status.
Time Frame: From date of inclusion until Radiographic progression, assessed up to 20 months
Population: There were an overall 40 patients with AR-V7 status known, 5 of them tested AR-V7 positive and 35 patients tested AR-V7 negative.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-label
Number analyzed (Participants) | 40
months
  AR-V7 negative: number analyzed (Participants) | 35
  AR-V7 negative | 5.53 [5.3 to 5.53]
  AR-V7 positive: number analyzed (Participants) | 5
  AR-V7 positive | 2.2 [0.3 to NA] — There were insufficient events, or insufficient follow-up, to estimate the upper limit of the confidence interval.

4. Secondary Outcome: Overall Survival (OS).
Time Frame: From date of inclusion until death from any cause or the last date the patient was known to be alive, assessed up to 20 months.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Open-label
Number analyzed (Participants) | 52
months | 14.8 [11.2 to NA] — Insufficient events or insufficient follow-up time, to estimate the upper limit of the confidence interval.

5. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE).
Description: Time to first SSE defined as the time from treatment initiation until SSE (pathological fractures, vertebral or non-vertebral, spinal cord compression, radiation or surgery to bone). For all other events, the start date of the event/medication/therapy was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From date of first drug administration until SSE, assessed up to 20 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-label
Number analyzed (Participants) | 52
months | NA [NA to NA] — The SSEs were reported in 5 patients (9.6%), therefore, the median time to first SSE was not reached

6. Secondary Outcome: Time to PSA Progression According to the ALSYMPCA Study Criteria.
Time Frame: From date of first study drug administration to when PSA progression is observed, assessed up to 20 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Open-label
Number analyzed (Participants) | 52
months | 3.3 [1.9 to NA] — Insufficient events or insufficient follow-up time, to estimate the upper limit of the confidence interval.

7. Secondary Outcome: PSA Progression
Description: PSA progression (defined as PSA elevation ≥ 25% and ≥ 2 ng/mL after 12 weeks).
Time Frame: From date of first study drug administration to when PSA progression is observed, assessed up to 20 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 52
Participants | 5

8. Secondary Outcome: Alkaline Phosphatase Level Response (AF), Normalization of Alkaline Phosphatase Level
Description: Progression defined as FA elevation ≥ 25% after 12 weeks
Time Frame: From date of first study drug administration until End of Treatment, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 52
Participants | 17

9. Secondary Outcome: Assessment of AR-V7 Mutation Evolution
Time Frame: From date of first study drug administration until End of Treatment, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 52
Participants
  Baseline Evaluation: AR-V7 Negative | 35
  Baseline Evaluation: AR-V7 Positive | 5
  Baseline Evaluation: Not reported | 12
  EoT evaluation: AR-V7 Negative | 26
  EoT evaluation: AR-V7 Positive | 1
  EoT evaluation: Not reported | 25

10. Secondary Outcome: Number of Participants With Change in CTCs Number
Description: CTC levels will be measured at the start and at the end of the study. Patients will be categorized based on their CTC levels: those with a CTC count higher than 5, lower than 5, and CTC not reported. A lower CTC count is considered a better outcome.
Time Frame: From date of first study drug administration until End of Treatment, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 52
Participants
  Baseline Evaluation: CTC ≥ 5 | 10
  Baseline Evaluation: CTC < 5 | 30
  Baseline Evaluation: CTC Not reported | 12
  EoT Evaluation: CTC ≥ 5 | 4
  EoT Evaluation: CTC < 5 | 24
  EoT Evaluation: CTC Not reported | 24

ADVERSE EVENTS:
Time Frame: Baseline up to 2 years after last dose.
Arm/Group | Open-label
All-Cause Mortality (participants affected / at risk) | 3/52
Serious Adverse Events (participants affected / at risk) | 11/52
Other Adverse Events (participants affected / at risk) | 30/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (N=52)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Uncontrolled pain (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Worsening general condition (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label (N=52)
Asthenia (General disorders) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Athralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
For several endpoints, the upper confidence interval could not be calculated because either 50% of patients at the endpoint were not reached (in the case of DFS) or were reached very late in the study, close to EoS (such as rPFS, OS and PSA) and we could not meaningfully state the value of this data due to lack of information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03002220/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03002220/SAP_001.pdf